CLINICAL TRIAL: NCT00265356
Title: The Impact of Positron Emission Tomography (PET) Imaging Prior to Liver Resection for Colorectal Adenocarcinoma Metastases: A Prospective, Multicentre Randomized Clinical Trial
Brief Title: Impact of Positron Emission Tomography Imaging Prior to Liver Resection for Colorectal Adenocarcinoma Metastases
Acronym: PETCAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CTA-Control-098389
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: Positron Emission Tomography (PET); Diagnostic Investigation; Colorectal cancer; Liver metastases; Liver surgery
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): PET diagnostic imaging
  Interventions: Procedure: PET diagnostic imaging
- 2 (No Intervention): No PET

INTERVENTIONS:
Procedure: PET diagnostic imaging — PET diagnostic imaging
  Other Names: Positron Emission Tomography
  Arms: 1

SUMMARY:
The purpose of this trial is to improve the management of patients with potentially surgically curable colorectal cancer liver metastases.

The primary objective is to determine the impact of pre-operative positron emission tomography (PET) on patients who have been assessed as having resectable colorectal cancer liver metastases by conventional imaging (computed tomography (CT) abdomen/thorax, colonoscopy), by determining the proportion of patients who have a change in management resulting from PET.

DETAILED DESCRIPTION:
Colorectal cancer remains a leading cause of death in men and women. A significant number of patients with colorectal cancer will either present with, or subsequently develop, liver metastases. In contrast to many other epithelial solid tumours, resection of colorectal cancer hepatic metastases results in long-term survival and even cure. However, despite state of the art CT imaging, 60-75% of patients who appear to have limited disease amenable to surgical resection will eventually die from extra-hepatic and recurrent hepatic metastases. If occult micrometastatic disease that becomes evident after liver resection could be detected reliably during pre-operative assessment, patients harboring more widespread disease could be spared a non-curative liver resection. This is one of the present challenges of liver surgery. PET imaging has the potential to improve the detection of both hepatic and extra-hepatic metastatic disease, not detected by conventional imaging modalities.

This prospective, multicenter trial will enroll patients with colorectal cancer liver metastases considered resectable, based on CT scans of the thorax, abdomen and pelvis, which demonstrate no evidence of extra-hepatic disease. A full colonoscopy within the preceding 12 months will ensure there is no local recurrence, or other primary cancer at the time of planned liver resection. These patients will be randomized to PET scan or not.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic proof of previous colorectal adenocarcinoma (not carcinoid, squamous cell cancer, gastrointestinal stromal tumor, or lymphoma)
2. Contrast-enhanced spiral CT scan of the thorax, and a tri-phasic CT scan of the abdomen and pelvis performed within 30 days (plus up to 14 days) before randomization demonstrating resectable metastasis(es) that are isolated to the liver
3. Full colonoscopy performed within the preceding 18 months showing no evidence of malignancy (other than a synchronous colorectal primary expected to be removed at time of liver resection)
4. Age over 18 years

Exclusion Criteria:

1. Extrahepatic disease including enlarged portal lymph nodes on CT
2. Prior liver resection
3. Previous radiofrequency ablation of malignant liver lesion
4. Systemic chemotherapy within three weeks prior to randomization
5. Radiotherapy within two months prior to randomization
6. Significant concurrent medical problems (e.g., uncontrolled diabetes, active cardiac disease, significant chronic obstructive pulmonary disease) making the patient unfit for surgery
7. Pregnant or lactating female
8. Unable to lie supine for imaging with PET
9. Previously treated cancer other than non-melanocytic skin cancer or carcinoma in situ of the cervix, unless disease-free for 5 years or greater
10. Patients who, at the time of the initial evaluation, have already undergone a whole body PET within 6 months prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2005-11; Primary Completion 2010-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
proportion of patients who have a change in management resulting from PET | 12 months

SECONDARY OUTCOMES:
proportion of patients precluded from having a liver resection because of additional metastatic disease identified on PET | 12 months
3-year overall survival of patients who undergo surgery with curative intent | 12 months
3-year overall survival of all patients | 12 months
sensitivity and specificity of PET in detecting other hepatic and extra-hepatic metastatic disease prior to a potentially curable liver resection for colorectal adenocarcinoma metastatic disease | 12 months
economic analysis of the addition of PET in the diagnostic work-up | 4 year
prognostic ability of the PET standard uptake value (SUV) in predicting 3-year overall survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven Gallinger, MD, Study Chair — University Health Network: Mount Sinai Hospital; Mark Levine, MD, Principal Investigator — Ontario Clinical Oncology Group (OCOG); Carol-anne Moulton, MD, Principal Investigator — University Health Network: Toronto General Hospital
Locations (9):
- Canada (9):
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Health Sciences, London, Ontario
  - The Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario

REFERENCES:
- [Derived] Serrano PE, Gafni A, Gu CS, Gulenchyn KY, Julian JA, Law C, Hendler AL, Moulton CA, Gallinger S, Levine MN. Positron Emission Tomography-Computed Tomography (PET-CT) Versus No PET-CT in the Management of Potentially Resectable Colorectal Cancer Liver Metastases: Cost Implications of a Randomized Controlled Trial. J Oncol Pract. 2016 Jul;12(7):e765-74. doi: 10.1200/JOP.2016.011676. Epub 2016 Jun 21. PMID 27328792
- [Derived] Moulton CA, Gu CS, Law CH, Tandan VR, Hart R, Quan D, Fairfull Smith RJ, Jalink DW, Husien M, Serrano PE, Hendler AL, Haider MA, Ruo L, Gulenchyn KY, Finch T, Julian JA, Levine MN, Gallinger S. Effect of PET before liver resection on surgical management for colorectal adenocarcinoma metastases: a randomized clinical trial. JAMA. 2014 May 14;311(18):1863-9. doi: 10.1001/jama.2014.3740. PMID 24825641